CLINICAL TRIAL: NCT06279806
Title: The Effect of Mobile Health Application Based on Transformational Learning Theory on Posttraumatic Growth in Women Diagnosed With Breast Cancer
Brief Title: The Effect of Mobile Health Application on Posttraumatic Growth in Women Diagnosed With Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Şengül Yaman Sözbir, Proffessor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SerapAlkas
Record Dates: First submitted 2024-02-04; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Posttraumatic Growth; Grief
Keywords: mobile health application; posttraumatic growth; grief; breast cancer; breast cancer survivor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: In order to ensure similarity between the groups, stratified block randomization will be used to assign the women in the sample group to the experimental and control groups. In this method, after stratification according to risk factors, block randomization is performed within each stratum. Since the type of treatment applied in breast cancer and marital status will significantly affect posttraumatic development, stratification was made in terms of these parameters. Stratum 1 in terms of treatment type: Mastectomy, 2nd stratum: Breast conserving surgery or reconstructive surgery during mastectomy; Stratum 1 in terms of partner presence: Has a partner, Stratum 2: No partner. In order to determine which stratum group the women who were found to meet the research criteria and who agreed to participate in the study were in, blocks will be formed with a combination of 4 and the assignment list will be determined through the www.randomizer.org website.
Who Masked: Outcomes Assessor
Masking Description: The data obtained from the research will be coded as A and B by an independent researcher and transferred to the SPSS program. The data will also be analyzed by an independent statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): Mobile health application use
  Interventions: Other: Mobile health application use
- Control Group (Experimental): Information of the breast cancer survivor period booklet
  Interventions: Other: Information of the breast cancer survivor period booklet

INTERVENTIONS:
Other: Mobile health application use — Women will be asked to use the app for at least 8 weeks. In order to monitor the usage, the researcher will monitor whether the women log in to the "Information and Counseling" section from the admin panel. Women who do not log in to the "Information and Counseling" section will be removed from the study at this stage. A weekly reminder will be sent to women via the mobile application. The questions asked by the participants through the question-and-answer section of the mobile health application will be examined every day and answered by the researcher between 10:00-11:00 every morning and 22:00-23:00 every evening. Likewise, the content shared by women in the forum section of the mobile application will be checked daily by the researcher and content that is harmful to women will be removed.
  Arms: İntervention Group
Other: Information of the breast cancer survivor period booklet — Women in the control group will be given information of the breast cancer survivor period booklet.
  Arms: Control Group

SUMMARY:
Breast cancer is the type of cancer that significantly affects women's health and causes the most mortal in women. Despite the high incidence of breast cancer, women living after breast cancer are increasing due to advances in early diagnosis and effective treatment options. Treatments are aimed at prolonging survival from breast cancer and enabling patients to live better. Women repeatedly experience many vital crises such as the diagnosis of cancer, the difficulties of the treatment process and the fear of recurrence in the post-treatment period. In the face of these crises, post-traumatic growth occurs when the individual's efforts to cope are transformed into positive psychological experiences. Positive experiences lead to improvement in women's life, while negative experiences make it difficult to cope and adapt. In order for post-traumatic growth to take place, women should be supported to cope with these negative emotions. The care given to patients during cancer treatment should be such as to support the change process that will help individuals adapt to the new lifestyle.This information and supportive care content should include the topics that women will need in the long term after the treatment, in addition to the diagnosis and treatment process. Generally, the education and counseling given to the patient at the last treatment appointment may be limited. Due to the long period from the last treatment appointment to the control appointment, patients cannot interact with healthcare professionals for a long time. Long-term side effects and needs of people may differ after breast cancer treatment. For this reason, the need for information and consultancy services of healthcare professionals continues in this process as well.Today, the use of remotely accessible mechanisms in the treatment of breast cancer and in the follow-up of women after treatment is increasing. It is thought that the mobile application to be developed within the scope of the project will increase the quality and efficiency of health services with an R&D and innovative approach and make these services accessible to everyone through digital technologies. In addition, our study will set an example for nursing care to be presented in one of the priority areas of health, such as cancer, through digital technologies. In our study, it is aimed to evaluate the effect of mobile health application based on Mezirow's Transformational Learning Theory on post-traumatic development in women with breast cancer. The research is a single center, parallel group, stratified block randomized controlled experimental study. It is planned to be conducted with 56 (intervention: 28, control: 28) women at Gazi University Health Research and Practice Center. The training content to be included in the mobile application has been determined by considering the results of the studies in the literature and the recommendations of international guides to determine the problems experienced by women with breast cancer during the post-treatment period. After receiving expert opinions on the subject content, the development process of the mobile application will be started. In the implementation phase of the study, the women in the intervention group will start using the mobile application 1 week after completing the active treatment chemotherapy and radiotherapy) process.The implementation of the study will last 8 weeks. At the end of eight weeks, data collection tools will be applied to the women. The final tests will be repeated 4 weeks after the end of the application. Starting from this period, women in the control group who want to use the application will also be included in the mobile application system. After completing the data collection tools, the analysis and reporting part will be started. Statistical analyzes will be made using SPSS Package Program (IBM SPSS Statistics 27). Student t test, Pearson Chi-square test, Independent Sample t test, Mann Whitney U test, One-Way Analysis of Variance or Friedman test will be used in the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Diagnosed with breast cancer Stage I-II-III-IV
* Having undergone breast cancer surgery
* To have completed cancer treatment,
* Being at the beginning of the remission period,
* Being able to read and write
* Having a cell phone with Android software

Exclusion Criteria:

* Having a diagnosed psychiatric illness,
* Receiving hormone therapy only,
* Having had any cancer before,
* Having a communication barrier (not speaking Turkish, speech/hearing impairment, etc.)
* Being visually impaired

Criteria for Exclusion from the Sample During the Study

* Not logging into the information and counseling panel of the mobile health application
* Wanting to leave study
* Failure to complete final tests
* Death of the participant

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-02-28 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Women's progression through the stages of grief | 12 week
  Mean scores on the Grief Psychological Reactions to Loss of Health Scale Psychological Reactions Scale due to Loss of Health: The scale has 30 items and is a 5-point Likert type (1: never, 5: always). The scale does not have a total score. Evaluation is made according to the scores obtained from the sub-dimensions. It is seen that as the score obtained from the sub-dimensions increases, there is an increase in the number of people experiencing each of the stages of grief. The scale has two different evaluations and two different subscale ratings.

SECONDARY OUTCOMES:
Women's increased level of posttraumatic development | 12 week
  Post-Traumatic Development Scale in Cancer Patients: The scale consists of 23 Likert-type scale items scored between 0-5. It is evaluated between "0" (I have never experienced it) and "5" (I have experienced it a lot). The lowest score to be obtained from the scale is 0, the highest score is 115, and the higher the score obtained from the scale, the more the individual develops after the trauma.